CLINICAL TRIAL: NCT02475356
Title: Special Drug Use Investigation of Mirena for Heavy Menstrual Bleeding and Dysmenorrhea
Brief Title: Prospective, Non-interventional, Multi-center Safety Study of Mirena for Heavy Menstrual Bleeding and Dysmenorrhea
Acronym: J-MIRAI
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18252
Record Dates: First submitted 2015-06-16; First posted 2015-06-18 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2020-12

CONDITIONS: Menorrhagia, Dysmenorrhea
Keywords: Mirena; Heavy Menstrual Bleeding; Dysmenorrhea; Japan; Post-marketing surveillance
MeSH Terms: conditions — Menorrhagia; Dysmenorrhea | interventions — Levonorgestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mirena: Mirena treatment group
  Interventions: Drug: Levonorgestrel IUS (Mirena, BAY86-5028)

INTERVENTIONS:
Drug: Levonorgestrel IUS (Mirena, BAY86-5028) — The treatment of Mirena should comply with the local product information.

SUMMARY:
The primary objective in this study is collecting post-marketing information on the safety. Thus, it includes information under the routine clinical practice on adverse events (AEs) and adverse drug reactions (ADRs) including expulsion and abnormal bleeding that occur within the first 12 months Mirena insertion.

The secondary objective(s) in this study is/are collecting information on Mirena effectiveness, such as periodic blood loss and Quality of life (QOL), use of analgesic and dysmenorrhea pain as far as these are recorded under routine clinical practice.

DETAILED DESCRIPTION:
This local, non-interventional, multicenter, single-cohort study using primary data includes patients treated with Mirena for Heavy menstrual bleeding(HMB) and/or dysmenorrhea (contraception is not included).

A total of 600 patients (valid for safety analysis) is planned to be enrolled in two years. No formal sample size estimation was conducted, it was determined based on feasibility.

Target population is patients with HMB and/or dysmenorrhea diagnosis. The treatment should be performed based on the product label in Japan. The standard observation period will last for 12 months from starting Mirena treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female patients diagnosed with HMB or/and dysmenorrhea.
* Patients for whom newly starting treatment with Mirena was made as per investigator's routine treatment practice
* Written informed consent

Exclusion Criteria:

* Patient whose purpose is only contraception

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female patients with Heavy menstrual bleeding (HMB) and/or dysmenorrhea in whom a decision to initiate treatment with Mirena has already been made will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 601 (Actual)
Dates: Start 2015-08-04 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse drug reaction | Up to 12 months
Number of participants with treatment-emergent adverse events (TEAEs) | Up to 12 months

SECONDARY OUTCOMES:
Change from baseline in bleeding characterized by Pictorial Blood loss Assessment Chart (PBAC) score to 12 months | Baseline and 12 months
Change from baseline in monthly bleeding intensities (the number of spotting and/or bleeding days) to 12 months | Baseline and 12 months
Change from baseline in Quality of Life parameters assessed using MMAS or MDQ score after 3 and 12 months | Baseline and 3 months, Baseline and 12 months
  MMAS: Menorrhagia Multi Attribute Score for Heavy Menstrual Bleeding and MDQ: Menstrual Distress Questionnaire for dysmenorrhea
Change from baseline in dysmenorrhea pain using Visual Analogue scale | Baseline and 1 month, Baseline and 3 months, Baseline and 6 months, Baseline and 12 months
Change from baseline in use of analgesics after Mirena insertion | Baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- [Derived] Momoeda M, Akira S, Harada T, Kitawaki J, Maeda N, Ota I, Yoshihara K, Takahashi N. Quality of Life of Japanese Dysmenorrhea/Heavy Menstrual Bleeding Patients Treated with Levonorgestrel Intrauterine Delivery System in a Real-World Setting. Adv Ther. 2022 Aug;39(8):3616-3634. doi: 10.1007/s12325-022-02205-2. Epub 2022 Jun 16. PMID 35705788